CLINICAL TRIAL: NCT05883579
Title: Application of Coronary Artery Chronic Total Occlusion (CTO) Scoring Systems Detecting Their Prediction Ability on CTO Percutaneous Coronary Intervention (PCI) Procedures
Brief Title: Application of Coronary Artery Chronic Total Occlusion Scoring Systems
Acronym: CTO-PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Khaled Saber Abdelaal Qayed, Principal investigator, Assiut University
Other Study IDs: CTO-PCI scores application
Record Dates: First submitted 2023-05-17; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Chronic Total Occlusion of Coronary Artery
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — doing percutaneous revascularization of chronic coronary total occlusion.

SUMMARY:
Studying the prediction ability of different CTO scoring systems on Asian CTO PCI population with their relation to technical success and developing a newer stepwise approach depending on these CTO scoring systems for choosing the suggested successful approach considering collateral channel assessment.

DETAILED DESCRIPTION:
Study of applying the Japenese CTO, Castle and Progress CTO scores on all coronary CTO PCI cohort done at national Taiwan university hospital (NTUH)

Study tools:

1. Basal demographic data collection( age, cardiovascular risk factors, patients clinical data, lesion characteristics, periprocedural complications).
2. The Japanese Chronic Total Occlusion (J-CTO) score calculated for assessment of CTO procedures complexity and predict the likelihood of guide wire crossing within 30 min, as assembled by Morino et al.

   The J-CTO score is the sum of the following 5 binary parameters: blunt proximal cap, calcification, bending >45°, length of occluded segment >20 mm, and previously failed PCI attempt. Each of these independent variables was assigned a value of 1 when present. With increasing probability of difficulty of wire crossing from 0 as easy till 5 as very difficult.
3. Also, the PROGRESS-CTO score calculated (reference website: https://www.progresscto.org/cto with evaluation of 4 baseline angiographic characteristics (proximal cap ambiguity, absence of retrograde collaterals, moderate or severe tortuosity, and LCX CTO) used to determine the likelihood of technical success with CTO PCI. Each of these independent variables was assigned a value of 1 when present. With increasing probability of difficulty of success from 0 as easy till 5 as very difficult.
4. Euro CTO CASTLE scoring calculation

   The CASTLE (coronary artery bypass graft history, age, stump anatomy, tortuosity degree, length of occlusion, and extent of calcification) model applied retrospectively on the patients with every item taking 1 point if present And Technical failure rates range from 8% (CASTLE score 0 to 1) to 35% (CASTLE score ≥4).
5. Collateral assessment including type (septal, epicardial or bypass grafts), size by Werner classification [is graded as: 0, no visible connection between the donor and the recipient coronary artery; 1, thread-like connection between the donor and the recipient coronary artery; 2, side-branch like connection between the donor and the recipient coronary artery], tortuosity degree as by the CC scoring system of the NTUH--> Channel tortuosity caculated as the presence of ≥2 high-frequency, successive curves (within 2 mm) in the context of epicardial collaterals and ≥1 high-frequency curve that failed to uncoil in diastole for septal channels (thus a measure of channel distensibility). A high-frequency curve is defined as a curve that is >180° occurring within a segment length <3× the diameter of the collateral.

And all these scores references and calculation items are mentioned in the references below….

ELIGIBILITY:
Inclusion Criteria:

* All coronary CTO PCI procedures done at national Taiwan university hospital (NTUH) with their data available for analysis from 2015 till the study data collection step.

Exclusion Criteria:

* Patients whom data not completed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: coronary CTO PCI patients done by experienced high volume operator at national Taiwan university hospital (NTUH) with their data available for analysis
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
comparison of the effecacy of using CTO scoring systems (J-CTO scoring, Castle Score and progress scoring along with the CC scoring in prediction of technical success. | Two months
  comaprling the three CTO scores for all CTO PCI patients done by experienced operator ( J-CTO scoring, Castle Score and progress scoring ) for prediction of technical success with higher scores indicating higher probability of difficulty along with the CC scoring in predicting higher chances of technical success in retrograde CTO PCI patients.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Rushdy, Professor, Study Chair — Assiut University; Paul Kao, Professor, Study Director — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Huang CC, Lee CK, Meng SW, Hung CS, Chen YH, Lin MS, Yeh CF, Kao HL. Collateral Channel Size and Tortuosity Predict Retrograde Percutaneous Coronary Intervention Success for Chronic Total Occlusion. Circ Cardiovasc Interv. 2018 Jan;11(1):e005124. doi: 10.1161/CIRCINTERVENTIONS.117.005124. PMID 29311284
- [Result] Werner GS, Ferrari M, Heinke S, Kuethe F, Surber R, Richartz BM, Figulla HR. Angiographic assessment of collateral connections in comparison with invasively determined collateral function in chronic coronary occlusions. Circulation. 2003 Apr 22;107(15):1972-7. doi: 10.1161/01.CIR.0000061953.72662.3A. Epub 2003 Mar 24. PMID 12665484
- [Result] Galassi AR, Werner GS, Boukhris M, Azzalini L, Mashayekhi K, Carlino M, Avran A, Konstantinidis NV, Grancini L, Bryniarski L, Garbo R, Bozinovic N, Gershlick AH, Rathore S, Di Mario C, Louvard Y, Reifart N, Sianos G. Percutaneous recanalisation of chronic total occlusions: 2019 consensus document from the EuroCTO Club. EuroIntervention. 2019 Jun 20;15(2):198-208. doi: 10.4244/EIJ-D-18-00826. PMID 30636678
- [Result] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Result] Tajti P, Burke MN, Karmpaliotis D, Alaswad K, Werner GS, Azzalini L, Carlino M, Patel M, Mashayekhi K, Egred M, Krestyaninov O, Khelimskii D, Nicholson WJ, Ungi I, Galassi AR, Banerjee S, Brilakis ES. Update in the Percutaneous Management of Coronary Chronic Total Occlusions. JACC Cardiovasc Interv. 2018 Apr 9;11(7):615-625. doi: 10.1016/j.jcin.2017.10.052. Epub 2018 Mar 14. PMID 29550088
- [Result] Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, Ochiai M, Noguchi Y, Kato K, Shibata Y, Hiasa Y, Doi O, Yamashita T, Hinohara T, Tanaka H, Mitsudo K; J-CTO Registry Investigators. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACC Cardiovasc Interv. 2011 Feb;4(2):213-21. doi: 10.1016/j.jcin.2010.09.024. PMID 21349461
- [Result] Galassi AR, Boukhris M, Azzarelli S, Castaing M, Marza F, Tomasello SD. Percutaneous Coronary Revascularization for Chronic Total Occlusions: A Novel Predictive Score of Technical Failure Using Advanced Technologies. JACC Cardiovasc Interv. 2016 May 9;9(9):911-22. doi: 10.1016/j.jcin.2016.01.036. Epub 2016 Apr 13. PMID 27085580
- [Result] Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, Alaswad K, Lombardi W, Grantham JA, Moses J, Christakopoulos G, Tarar MNJ, Rangan BV, Lembo N, Garcia S, Cipher D, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016 Jan 11;9(1):1-9. doi: 10.1016/j.jcin.2015.09.022. PMID 26762904
- [Result] Szijgyarto Z, Rampat R, Werner GS, Ho C, Reifart N, Lefevre T, Louvard Y, Avran A, Kambis M, Buettner HJ, Di Mario C, Gershlick A, Escaned J, Sianos G, Galassi A, Garbo R, Goktekin O, Meyer-Gessner M, Lauer B, Elhadad S, Bufe A, Boudou N, Sievert H, Martin-Yuste V, Thuesen L, Erglis A, Christiansen E, Spratt J, Bryniarski L, Clayton T, Hildick-Smith D. Derivation and Validation of a Chronic Total Coronary Occlusion Intervention Procedural Success Score From the 20,000-Patient EuroCTO Registry: The EuroCTO (CASTLE) Score. JACC Cardiovasc Interv. 2019 Feb 25;12(4):335-342. doi: 10.1016/j.jcin.2018.11.020. Epub 2019 Jan 30. PMID 30711551
- [Result] Ellis SG, Burke MN, Murad MB, Graham JJ, Badawi R, Toma C, Meltser H, Nair R, Buller C, Whitlow PL; CAPS Group. Predictors of Successful Hybrid-Approach Chronic Total Coronary Artery Occlusion Stenting: An Improved Model With Novel Correlates. JACC Cardiovasc Interv. 2017 Jun 12;10(11):1089-1098. doi: 10.1016/j.jcin.2017.03.016. PMID 28595879
- [Result] Li Y, Xu N, Zhang J, Li M, Lu Z, Wei M, Lu B, Zhang Y. Procedural success of CTO recanalization: Comparison of the J-CTO score determined by coronary CT angiography to invasive angiography. J Cardiovasc Comput Tomogr. 2015 Nov-Dec;9(6):578-84. doi: 10.1016/j.jcct.2015.07.005. Epub 2015 Jul 23. PMID 26232276
- [Result] Salinas P, Gonzalo N, Moreno VH, Fuentes M, Santos-Martinez S, Fernandez-Diaz JA, Amat-Santos IJ, Ojeda FB, Borrego JC, Cuesta J, Hernandez JMT, Diego-Nieto A, Dubois D, Galeote G, Goicolea J, Gutierrez A, Jimenez-Fernandez M, Jimenez-Mazuecos J, Jurado A, Lacunza J, Lee DH, Lopez M, Lozano F, Martin-Moreiras J, Martin-Yuste V, Millan R, Minana G, Mohandes M, Morales-Ponce FJ, Nunez J, Ojeda S, Pan M, Rivero F, Robles J, Rodriguez-Leiras S, Rojas S, Rondan J, Rumiz E, Sabate M, Sanchis J, Vaquerizo B, Escaned J. Choice of CTO scores to predict procedural success in clinical practice. A comparison of 4 different CTO PCI scores in a comprehensive national registry including expert and learning CTO operators. PLoS One. 2021 Apr 2;16(4):e0245898. doi: 10.1371/journal.pone.0245898. eCollection 2021. PMID 33798205
- [Result] Kalogeropoulos AS, Alsanjari O, Keeble TR, Tang KH, Konstantinou K, Katsikis A, Jagathesan R, Aggarwal RK, Clesham GJ, Kelly PA, Werner GS, Hildick-Smith D, Davies JR, Karamasis G. CASTLE score versus J-CTO score for the prediction of technical success in chronic total occlusion percutaneous revascularisation. EuroIntervention. 2020 Apr 3;15(18):e1615-e1623. doi: 10.4244/EIJ-D-19-00352. PMID 31270036